CLINICAL TRIAL: NCT00276393
Title: Randomized Trial Comparing Insulin Glargine to Ultra-Lente Insulin in Type I Diabetes
Brief Title: Treatment Trial Evaluating Long Acting Insulin in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 70-02; 1A4372
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: Basal insulin

SUMMARY:
Patients with type 1 diabetes trained in multiple daily insulin injection were treated with two diffferent kinds of long acting insulin preparations. The two insulin preparations were glargine and ultralente insulin. Patients were randomized to receive one of the two insulin preparations for the first 4 months followed by the second preparation for a further four months. Short acting insulin used was the same during both periods. We found that glargine insulin was better than ultralente insulin in our study.

DETAILED DESCRIPTION:
Multiple daily insulin injection (MDI) programs are commonly accompanied by considerable glycemic variation and hypoglycemia. In order to determine whether use of insulin glargine as a basal insulin would result in comparable HbA1c with less glycemic variation and hypoglycemia than ultralente insulin, 22 individuals with type 1 diabetes, experienced with MDI, and a HbA1c of <7.8 % were randomized, to receive either glargine or ultralente as the basal insulin for 4-months. Aspart insulin was used as the prandial. Physicians providing insulin dose adjustment advice were masked to the type of basal insulin. Treatment with glargine resulted in lower mean HbA1c, less nocturnal variability , and less hypoglycemia primarily due to less daytime hypoglycemia (p=0.002). On the other hand, serious hypoglycemia and average glucose concentration measured with continuous glucose monitoring system (CGMS) did not differ. We conclude that, while use of either ultralente or glargine as a basal insulin can result in excellent glycemic control, treatment with glargine is associated with slightly but significantly lower HbA1C, with less nocturnal glycemic variability and less hypoglycemia.

ELIGIBILITY:
Type 1 diabetes, HbA1c < 7.8%, who have had prior instruction in a complex insulin program, and presently using a MDI insulin program with basal insulin preparations of Glargine or Ultralente and Humalog as the short acting insulin, should be free of hepatorenal abnormalities and hypoglycemia unawareness; non-pregnant, and should be able to perform frequent self monitoring of blood glucose (SMBG) and accept the use of continuous glucose monitoring system (CGMS). They should also possess the skill and understanding of insulin dose adjustments and supplementation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2002-07; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
HbA1c
Hypoglycemic events
Nocturnal hypoglycemia
Mean glucose
Mean fasting glucose

SECONDARY OUTCOMES:
Days of titration of basal insulin
Fear of hypoglycemia
Continuos glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Yogish C. Kudva, M.B.B.S, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Kudva YC, Basu A, Jenkins GD, Pons GM, Quandt LL, Gebel JA, Vogelsang DA, Smith SA, Rizza RA, Isley WL. Randomized controlled clinical trial of glargine versus ultralente insulin in the treatment of type 1 diabetes. Diabetes Care. 2005 Jan;28(1):10-4. doi: 10.2337/diacare.28.1.10. PMID 15616226